CLINICAL TRIAL: NCT02757313
Title: Neuroscience of Marijuana Impaired Driving
Acronym: MJDriving
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Hartford Hospital (Other); National Institute on Drug Abuse (NIDA) (NIH); Montana State University (Other); Maastricht University (Other); The Mind Research Network (Other)
Responsible Party: Principal Investigator, Godfrey Pearlson, Founding Director Olin Neuropsychiatry Research Center; Professor Yale University, Yale University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Other
Other Study IDs: 1507016175; 1R01DA038807-01A1 (NIH)
Record Dates: First submitted 2016-04-11; First posted 2016-05-02 (Estimated); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Marijuana Impairment
Keywords: marijuana; driving; THC; cannabis; intoxication; MRI
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol; nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regular Users (Experimental): People who use marijuana regularly will be given a low dose THC marijuana, high dose THC marijuana and placebo marijuana, in a randomized order, at the study visits.
  Interventions: Drug: Low dose THC marijuana; Drug: High dose THC marijuana; Drug: Placebo marijuana
- Occasional Users (Experimental): People who use marijuana occasionally will be given a low dose THC marijuana, high dose THC marijuana and placebo marijuana, in a randomized order, at the study visits.
  Interventions: Drug: Low dose THC marijuana; Drug: High dose THC marijuana; Drug: Placebo marijuana

INTERVENTIONS:
Drug: Low dose THC marijuana
  Other Names: THC, cannabis
Drug: High dose THC marijuana
  Other Names: THC, cannabis
Drug: Placebo marijuana
  Other Names: THC, cannabis

SUMMARY:
Marijuana is one of the most widely used substances. However, marijuana intoxication is not fully understood in relation to driving. This study will help the investigators learn more about the potential impairments related to marijuana intoxicated driving. A combination of MRI and neuropsychological tests (which are computer and paper/pencil tasks) will be used to measure intoxication and impairment. This study will also assess levels of marijuana in blood and saliva samples. This study takes place in Hartford, Connecticut.

DETAILED DESCRIPTION:
Cannabis is a commonly abused drug whose use cuts across social class, is linked to cognitive impairment, and may be a major contributor to intoxication-related accidents - either alone or with alcohol. However, cannabis intoxication is little studied in relation to driving compared to alcohol. Not only does the current NHTSA Strategic Plan for Behavioral Research prioritize understanding how drugs other than alcohol contribute to traffic crashes, it has recently become more pressing to understand the effects of cannabis because of increasing rates of legalized medical and/or recreational use, that will likely result in more cannabis intoxicated drivers. Social and legal policy will be unable to effectively address the many concerns about driving safety raised by more frequent and widespread use of cannabis without new research to better determine the parameters within which cannabis use does, or does not, increase automobile accident risk. The purpose of this study is to better describe specific, driving-related cognitive impairments caused by acute cannabis intoxication, their persistence over time, underlying functional brain anatomy, and relationship to performance on a state-of the art validated simulated driving task in which the investigators have prior experience. In a randomized, counterbalanced, double-blinded fashion, the investigators will administer two cannabis doses and placebo of smoked cannabis (paced inhalation using a vaporizer) to 48 regular cannabis users and 48 occasional cannabis users on 3 separate occasions. Following cannabis dosing cognitive and driving impairment will be assessed longitudinally for several hours using a combination of fMRI and neuropsychological tests, to clarify relationships between subjective and objective measures of intoxication and of impairment, that include expert assessment of THC and its metabolite levels in blood and saliva. This study takes place in Hartford, Connecticut.

ELIGIBILITY:
Inclusion Criteria:

* Must have a current driver's license
* Have used marijuana before
* Right handed

Exclusion Criteria:

* Females who are pregnant or breast feeding
* Unable or unsafe to have an MRI
* Any serious medical, or neurological disorder
* Any psychiatric disorder
* No major head traumas

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2016-10; Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Change in performance on fMRI simulated driving Gap Acceptance Task | Post drug administration at: 30 min, 3 hours and 5.25 hours
  The Gap Acceptance Task measures strategic control of the vehicle. Strategic control of the vehicle is measured by size of headway gaps that the participant chooses in pulling out into a stream of traffic.
Change in performance on fMRI simulated driving Road Tracking Task. | Post drug administration at: 30 min, 3 hours and 5.25 hours
  The Road Tracking Task measures operational control of the vehicle. Operational control is measured by standard deviation of lane position from the center point of the lane.
Change in performance on fMRI simulated driving Car Following Task. | Post drug administration at: 30 min, 3 hours and 5.25 hours
  The Car Following Task measures tactical control of the vehicle. Tactical control of the vehicle is measured by following distance from a lead vehicle.
Change in concentration of THC/metabolites in oral fluid tested using Draeger Drug Detection Kits | Baseline and post drug administration at: 5 min, 20 min, 1 hr 10 min, 1 hr 45 min, 2 hrs 30 min, 4 hrs, and 6 hrs 30 min,
  Saliva samples will be taken at 8 total time points throughout the day using the Draeger Drug Detection kits to assess for changes in concentration of THC and its metabolites.
Change in concentration of THC/metabolites in oral fluid tested using Quantisal Oral Fluid Collection devices. | Baseline and post drug administration at: 5 min, 20 min, 1 hr 10 min, 1 hr 45 min, 2 hrs 30 min, 4 hrs, and 6 hrs 30 min,
  Saliva samples will be taken at 8 total time points throughout the day using the Quantisal Oral Fluid Collection devices to assess for changes in concentration of THC and its metabolites.
Change in concentration of THC/metabolites in blood samples. | Baseline and post drug administration at: 5 min, 20 min, 1 hr 10 min, 1 hr 45 min, 2 hrs 30 min, 4 hrs, and 6 hrs 30 min,
  Blood samples will be taken at 8 total time points throughout the day to assess for changes in concentration of THC and its metabolites.
Marijuana performance changes on the Critical Tracking Task. | Post drug administration at two of the following time points (which varies dependent on the visit day): 2 hours; 4.25 hours; 6.5 hours
  The Critical Tracking Task assesses visuomotor tracking, it will be administered prior to dosing and at various time points after dosing.
Marijuana performance changes on the Tower of London task. | Post drug administration at two of the following time points (which varies dependent on the visit day): 2 hours; 4.25 hours; 6.5 hours
  The Tower of London is a task that assesses executive functioning, it will be administered prior to dosing and at various time points after dosing.
Marijuana performance changes on the Cogstate 1-back/2-back task. | Post drug administration at two of the following time points (which varies dependent on the visit day): 2 hours; 4.25 hours; 6.5 hours
  The Cogstate 1-back/2-back task assesses working memory, it will be administered prior to dosing and at various time points after dosing.
Marijuana performance changes on the Cogstate Detection Task. | Post drug administration at two of the following time points (which varies dependent on the visit day): 2 hours; 4.25 hours; 6.5 hours
  The Cogstate Detection Task assesses processing speed, it will be administered prior to dosing and at various time points after dosing.
Marijuana performance changes on the Cogstate Set Shifting Task. | Post drug administration at two of the following time points (which varies dependent on the visit day): 2 hours; 4.25 hours; 6.5 hours
  The Cogstate Set Shifting Task assesses executive functioning, it will be administered prior to dosing and at various time points after dosing.

SECONDARY OUTCOMES:
Change in performance on fMRI Set-Shifting paradigm. | Post drug administration at: 1.25 hours, 3.5 hours and 6 hours
  The set shifting paradigm measures attentional and executive domains.
Change in performance on fMRI Time Estimation paradigm. | Post drug administration at: 1.25 hours, 3.5 hours and 6 hours
  The time estimation paradigm measures misjudgment of time intervals based on participant responses indicating whether one time interval was the same, longer or shorter than the previous time interval.

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey Pearlson, Principal Investigator — Founding Director Olin Research Center; Professor Yale University
Locations (1):
- Olin Neuropsychiatry Research Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No